CLINICAL TRIAL: NCT03656549
Title: Individualized Pemetrexed Dosing in Patients With Non-small Cell Lung Cancer or Mesothelioma Based on Renal Function to Improve Treatment Response
Brief Title: Dose Individualization of Pemetrexed - IMPROVE-I
Acronym: IMPROVE-I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPROVE-I
Record Dates: First submitted 2018-05-14; First posted 2018-09-04 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer; Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma | interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impaired renal function (Experimental): patients will be treated with pemetrexed, with dosing based on renal function in combination with oral folinic acid rescue
  Interventions: Drug: Pemetrexed + oral folinic acid rescue

INTERVENTIONS:
Drug: Pemetrexed + oral folinic acid rescue — 3+3 dose escalation study of pemetrexed in patients with impaired renal function in combination with roal folinic acid rescue

SUMMARY:
Rationale:

Pemetrexed is a multi-targeted folate antagonist, which is primarily indicated for the treatment of advanced non-small cell lung cancer (NSCLC) and mesothelioma. Dosing of cytotoxic agents like pemetrexed requires balancing the dual risk of sub-therapy and toxicity. Administration of pemetrexed to patients with a creatinine clearance <45 ml/min is currently not advised. Pemetrexed is dosed based on body surface area (BSA), while renal function and dose are the sole determinants for systemic exposure. This causes these issues:

1. In patients with renal dysfunction, BSA-based dosing may lead to haematological toxicity
2. Patients have to discontinue treatment due to declining renal function, and are withheld effective treatment

Objective:

The main objective is to develop a safe dosing regimen for pemetrexed in patients with renal impairment.

Study design:

IMPROVE-I is a single arm dose finding study to assess the feasibility of renal function-based dosing of pemetrexed in combination with folinic acid or folinic acid and pegfilgrastim in renally impaired patients.

Study population:

IMPROVE-I includes a maximum of twelve evaluable patients with NSCLC or mesothelioma with a renal function <45ml/min that meet all other requirements for pemetrexed treatment.

Intervention:

IMPROVE-I: patients who have an indication for treatment with pemetrexed, but who have an impaired renal function will be treated with pemetrexed in combination with folinic acid rescue therapy. Dosing of pemetrexed will be based on renal function to reach the target AUC. As a safety measure a minimum of 4 intra-patient dose escalations in the first patient will be performed starting from 10% of the target AUC. A standard 3+3 study design is used. If folinic acid is not sufficient to prevent haematotoxicity, prophylactic treatment with pegfilgrastim will be added to the combination therapy.

Main study endpoints:

IMPROVE-I: The fraction of patients safely reaching the target dose.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

We consider the extra burden from participating in the planned studies limited. The extra interventions compared to routine care, consist of sampling extra blood. The pharmacokinetic assessments require placement of one additional intravenous catheter. To ensure minimal impact of study participation on daily life, we will use a limited sampling strategy. Patients may benefit from participating in IMPROVE I, as they will be treated with a potentially safe and effective drug that is dosed individually, which prevents toxic exposure.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Eligible for treatment with pemetrexed-based chemotherapy based on indication
3. Estimated creatinine clearance <45ml/min
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
5. Subject is able and willing to sign the Informed Consent Form

Exclusion Criteria:

1. Conditions that affect haemostasis in a way that blood drawing is complicated (to be assessed by physician)
2. Contraindications for treatment with pemetrexed in line with the summary of product characteristics (SmPC) (except for creatinine clearance <45 ml/min in IMPROVE-I)

   1. Hypersensitivity to the active substance or to any of the excipients
   2. Pregnancy or lactation
   3. Concomitant yellow fever vaccine
3. The presence of clinically relevant pharmacokinetic interactions, according to the current SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
The fraction of patients safely reaching the target dose in combination with folinic acid or folinic acid and G-CSF, with the target dose being the dose most likely to result in an AUC of 164 mg*h/L. | 3 months

SECONDARY OUTCOMES:
The AUC of pemetrexed for each patient at 100% dose | 3 months
  mg*h/L
Complete blood count prior to start of every cycle and on day 7 and 14 after administration | From start of treatment to the last day of the 4th cycle of chemotherapy
The incidence of hematologic dose limiting toxicities (DLT) and adverse events, as measured with the CTCAE V4' | 3 months
  through listing
The incidence of non-hematologic dose limiting toxicities (DLT) and adverse events, as measured with the CTCAE V4 | 3 months
  through listing
The incidence of toxicity-related dose reductions, treatment delays and treatment discontinuation | 3 months
  through listing

CONTACTS AND LOCATIONS:
Overall Officials: Rob ter Heine, PhD, Principal Investigator — Radboud University Medical Center
Locations (6):
- Netherlands (6):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Antoni van Leeuwenhoek, Amsterdam
  - Catharina hospital, Eindhoven
  - Maastricht University Medical centre, Maastricht
  - Radboud university medical centre, Nijmegen
  - Erasmus University Medical Centre, Rotterdam

REFERENCES:
- [Derived] de Rouw N, de Boer M, Boosman RJ, van den Heuvel MM, Burger DM, Lieverse JE, Derijks HJ, Frederix GWJ, Ter Heine R. The Pharmacoeconomic Benefits of Pemetrexed Dose Individualization in Patients With Lung Cancer. Clin Pharmacol Ther. 2022 May;111(5):1103-1110. doi: 10.1002/cpt.2529. Epub 2022 Feb 21. PMID 35048355
- [Derived] Boosman RJ, Dorlo TPC, de Rouw N, Burgers JA, Dingemans AC, van den Heuvel MM, Hendriks LEL, Biesma B, Aerts JGJV, Croes S, Mathijssen RHJ, Huitema ADR, Ter Heine R. Toxicity of pemetrexed during renal impairment explained-Implications for safe treatment. Int J Cancer. 2021 Oct 15;149(8):1576-1584. doi: 10.1002/ijc.33721. Epub 2021 Jul 7. PMID 34181276